CLINICAL TRIAL: NCT04584606
Title: Ain Shams University Experience: Clinical Characteristics and Outcome Determinants of Hospitalized Covid-19 Patients at Ain Shams University Obour Hospital
Brief Title: Ain Shams University Experience: Clinical Determinants of Hospitalized COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf A Elmaraghy, Assistant Professor, Ain Shams University
Other Study IDs: FMASU P30/ 2020
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lab workup (on admission and regularly during follow up). — Complete blood count with differential leucocytic count. Absolute lymphocytic and neutrophilic count. Liver functions: Aspartate transaminase and Alanine transaminase . Renal functions: Blood urea nitrogen, serum Creatinine. HbA1C. C-reactive protein (quantitative). Serum ferritin level. D - dimer level (quantitative). Coagulation profile (Prothrombin time/ Partial thromboplastin time/ International normalized ratio).
  Troponin level. Arterial blood gases when needed.
  Other Names: culture, imaging

SUMMARY:
COVID-19 as a novel disease, different disease patterns were observed worldwide, and many treatment plans were tried. So, it is important to investigate the Egyptian clinical characteristics and different factors that determine the patient's 'outcome

DETAILED DESCRIPTION:
Investigators will convey the Ain Shams University experience as the first university in Egypt to designate one of its hospitals (Ain Shams University Obour Hospital) for management of confirmed COVID19 cases. investigators will try to identify the characteristics of the disease as regards the clinical, laboratory and imaging abnormalities and to assess the outcome determinants. It is a retrospective observational cohort study at Ain Shams University Obour Hospital. All adult patients from both sexes with positive nucleic acid testing for severe adult respiratory syndrome Coronavirus (SARS-CoV-2)will be included.

Clinical criteria, laboratory data, radiological findings, hospital course and patient outcome will be anonymously collected from records.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients from both sexes with positive nucleic acid testing for severe adult respiratory syndrome Coronavirus (SARS-CoV-2).
* Standard of care arm of the ongoing clinical trials will be included in our study.

Exclusion Criteria:

* mild cases who don't need hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) patients from both sexes with positive nucleic acid testing for severe adult respiratory syndrome Coronavirus (SARS-CoV-2).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Recovery | Until patient is discharged or up to 12 weeks whichever comes first
  Recovery defined as resolution of fever without the use of antipyretics, improvement of respiratory symptoms (e.g., cough, dyspnea) and no need for supplemental oxygen
Mortality | Until patient is discharged or up to 12 weeks whichever comes first
  All cause mortality

SECONDARY OUTCOMES:
Conversion of nucleic acid testing for SARS-CoV-2 from positive to negative. | Until patient is discharged or up to 12 weeks whichever comes first
  Detected by Polymerase Chain Reaction (PCR) test for nasopharyngeal swab
Radiological progression of the COVID 19 disease | Until patient is discharged or up to 12 weeks whichever comes first
  detected by measuring the extent of pulmonary lesion in high resolution computed tomography (HRCT) of the chest
Functional progression of the COVID 19 disease | Until patient is discharged or up to 12 weeks whichever comes first
  increase oxygen demands detected by arterial blood gases analysis and/or pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Elmaraghy, Principal Investigator — Ain Shams University, Faculty of Medicine
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: Undecided